CLINICAL TRIAL: NCT03005561
Title: Multi Center, Interventional, Randomized Study Detection of Difficulties and Improvement Compliance to Growth Hormone Treatment
Brief Title: Detection of Difficulties and Improvement Compliance to Growth Hormone Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Eli Hershkovitz (Other)
Responsible Party: Sponsor-Investigator, Prof. Eli Hershkovitz, Prof., Soroka University Medical Center
Organization: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0223-16sor
Record Dates: First submitted 2016-12-19; First posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Growth Hormone Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): 100 participants that will be participating in the Play Back meetings.
  Interventions: Behavioral: Play Back Sessions
- Control (No Intervention): 100 participants that will not be participating in the Play Back meetings.

INTERVENTIONS:
Behavioral: Play Back Sessions — 100 participants that will be participating in two Play Back meetings. Playback define that improvisation as a theater facilitator asks the audience to share moments, feelings and stories of his daily life, and a group of actors improvise their stories in front of the stage as a kind of "play-back". Unlike hobbies such as sports or singing, the method allows not only to unload the tensions but also communication and collaboration. It is very reminiscent of psychodrama, but unlike, is not considered a therapeutic tool.
  Arms: Intervention

SUMMARY:
In the last 50 years the use of growth hormone (rhGH, somatropin) has become commonly to treat problems such as GH deficiency, chronic renal failure and Turner syndrome and Prader-Willi. Giving the hormone in childhood and adolescence is designed to accelerate growth to close the gap in the average population and reach a final height is normal, while minimizing risks and costs.

Noncompliance to treatment with GH is common; Other estimates are that one third to one half of patients do not comply with the provisions as require. This may result in linear growth depreciation, unnecessary diagnostic tests, unnecessary change of dosage and treatment and higher costs.

Many studies have been devoted to locating factors make it difficult to adhere to their chronic diseases in children, including conditions that require treatment with GH.

Pain is the primary cause for difficulties. In recent decades, many resources were devoted to research and development of ways of dealing with pain in all aspects.

In order to implement all of the information collected, appropriate interventions medium should be found; In this study we intend to use the method of playback. Playback define that improvisation as a theater facilitator asks the audience to share moments, feelings and stories of his daily life, and a group of actors improvise their stories in front of the stage as a kind of "play-back". Unlike hobbies such as sports or singing, the method allows not only to unload the tensions but also communication and collaboration. It is very reminiscent of psychodrama, but unlike, is not considered a therapeutic tool.

Assumption:

Intervention of two playback meetings during the year will uncover the difficulties and engage ways of dealing with pain. That will reduce the difficulties caused by GH injections and improve compliance to treatment.

DETAILED DESCRIPTION:
In the last 50 years the use of growth hormone (rhGH, somatropin) has become commonly to treat problems such as GH deficiency, chronic renal failure and Turner syndrome and Prader-Willi. Giving the hormone in childhood and adolescence is designed to accelerate growth to close the gap in the average population and reach a final height is normal, while minimizing risks and costs.

Noncompliance to treatment with GH is common; Other estimates are that one third to one half of patients do not comply with the provisions as require. This may result in linear growth depreciation, unnecessary diagnostic tests, unnecessary change of dosage and treatment and higher costs.

GH therapy in all non-yielding satisfactory results, it is recommended first of all to consider noncompliance before turning to look for other causes.

Many studies have been devoted to locating factors make it difficult to adhere to their chronic diseases in children, including conditions that require treatment with GH.

Pain is the primary cause for difficulties. Despite the pain seems fairly simple phenomenon, it is actually very complex. Untreated pain is manifested prominently course and immediate distress to the child and the parent, but it has other deep effects; It seems that pain not receiving treatment at early stages in children's lives adversely affects the central nervous system development. This assumption is supported by various studies.

Pain is a force in shaping behavior; In recent decades, many resources were devoted to research and development of ways of dealing with pain in all aspects.

In order to implement all of the information collected, appropriate interventions medium should be found; In this study we intend to use the method of playback. Playback define that improvisation as a theater facilitator asks the audience to share moments, feelings and stories of his daily life, and a group of actors improvise their stories in front of the stage as a kind of "play-back". Unlike hobbies such as sports or singing, the method allows not only to unload the tensions but also communication and collaboration. It is very reminiscent of psychodrama, but unlike, is not considered a therapeutic tool.

Assumption:

Intervention of two playback meetings during the year will uncover the difficulties and engage ways of dealing with pain. That will reduce the difficulties caused by GH injections and improve compliance to treatment.

Study Population:

1. This is a pilot study in with a total of 200 participants treated with GH therapy.
2. Intervention group - 100 participants that will be participating in the Play Back meetings.
3. Control group - 100 participants with similar demographic s that will not participate in the play back meetings.

Patients will be divided randomly into groups. The following data will be collected-

* Height (SDS)
* Growth rate (SDS)
* IGF-1 (by SDS) - a sample taken on the first visit (time 0 and the last visit six months later).
* Accountability - empty ampoules of growth hormone (collected on a visit to No. 3 - After three months and the last visit, after six months).

Inclusion criteria:

1. Patients diagnosed with a growth hormone deficiency
2. Patients treated with growth hormone for at least two years.
3. The patient and parent signing an inform consent in the mother tongue.
4. Patients speakers and readers of Hebrew.
5. Age range: Boys 7 years to 12 years, Girls 7 years to 11 years.

Exclusion criteria:

1. Patients receiving growth hormone for other reasons.
2. Patients with comorbidities (celiac disease, hypothyroidism).
3. Children who began signs of puberty (Tanner 2 or higher).
4. Patients who completed growth, closed epiphysis.

The information collected in the study will be typed in encoder. The list that links the subject and the code given to them will be kept in the ISF, that will be be accessible only to the study team. The questionnaires of the participants will be identified through a personal code given to each of the participants and will be stored in a dedicated research folder in the Endocrinology and diabetes at Soroka Medical Center.

The intervention protocol:

Visit no.1:

1. Parents and patient will sign the ICF.
2. Patients will be randomized.
3. Height and Weight will be measured.
4. Patient / parent will answer questionnaires regarding their compliance to GH treatment, their difficulties and the way the deal with pain - if patient is below age of 8, his parent will complete the questionnaire.
5. IGF-1 blood sample will be collected.
6. Patients and parents will be guided to bring their empty ampoules for the next study visit and also to the last visit.
7. Patients that randomized to the intervention group will meet the Play Back team for the first session.

Visit no.2:

This visit will take place one month after the first visit. Patients that randomized to the intervention group will meet the Play Back team for the first session.

The meeting will be divided for 2 age groups: the first for 7-9 years old participants, and the second one for 10-12 years old participants.

Visit no.3:

This visit will take place 3 months after the first visit. Patients that randomized to the intervention group will meet the Play Back team for the second session.

Visit no.4:

This visit will take place 6 months after the first visit.

1. Height and Weight will be measured.
2. IGF-1 blood sample will be collected.
3. Patient / parent will answer questionnaires regarding their compliance to GH treatment, their difficulties and the way the deal with pain - if patient is below age of 8, his parent will complete the questionnaire.
4. Drug accountability. System analysis and processing results Descriptive statistics quantitative variables (such as age)that distribute normally are shown as averages ± SD. Quantitative variables that do not show normal distribution (the number of days of hospitalization) will be presented as median values between quarterly domain. Categorical variables (such as gender) will be out of proportion.

Univariate analyzes

Comparison of different variables between groups will be carried out according to the following rules:

Quantitative variables (such as age)that distribute normally will be compared using the t test for independent samples.

Variables that do not show normal distribution as the number of days of hospitalization between the two groups will be compared using the Mann-Whitney test. Categorical variables such as sex, will be compared using the chi-squared test.

Analysis of correlations between different variables will be using Pearson and Spearman correlations based on the distribution and type of data.

Weight and height data IGFI will be compared between subgroups according to a change in HtSDS since the start of growth hormone therapy to baseline.

A multivariate model Checking the compliance level logistic regression model was constructed multivariate where the dependent variable will be high responsiveness and low responsiveness dichotomous variable (if the patient has more than 80% response variable will receive the 1 or not (less than 80%) then receives a value of 0). Independent variables will be different risk factors which have passed the initial data analysis phase.

All statistical tests of significance level will alpha = 0.05 two-sided unless stated otherwise. All pv values shall be rounded to two decimal places.

Data analysis will be performed in Microsoft SPSS version 22.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with a growth hormone deficiency
2. Patients treated with growth hormone for at least two years.
3. The patient and parent signing an inform consent in the mother tongue.
4. Patients speakers and readers of Hebrew.
5. Age range: Boys 7 years to 12 years, Girls 7 years to 11 years.

Exclusion Criteria:

1. Patients receiving growth hormone for other reasons.
2. Patients with comorbidities (celiac disease, hypothyroidism).
3. Children who began signs of puberty (Tanner 2 or higher).
4. Patients who completed growth, closed epiphysis.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change in height | 6 months
  change in height between visit no.1 and last visit.

SECONDARY OUTCOMES:
Change in weight | 6 months
  change in weight between visit no.1 and last visit.

OTHER OUTCOMES:
Change in IGF-1 | 6 months
  change in IGF-1 between visit no.1 and last visit.

IPD SHARING:
Plan to Share IPD: Undecided